CLINICAL TRIAL: NCT01026779
Title: Rotavirus Gastroenteritis and Vaccine Usage in Rhode Island: Active Hospital-Based Surveillance, Serotype Surveillance and a Case-Control Study
Brief Title: Rotavirus Gastroenteritis and Vaccine Usage in Rhode Island
Status: Completed | Type: Observational
Sponsor: Lifespan (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Penelope H. Dennehy, Principal Investigator, Lifespan
Other Study IDs: HCH-001
Record Dates: First submitted 2009-12-02; First posted 2009-12-04 (Estimated); Last update posted 2019-11-14 (Actual); Status verified 2019-11

CONDITIONS: Rotavirus Gastroenteritis
Keywords: rotavirus; gastroenteritis; vaccine; case-control study; serotype
MeSH Terms: conditions — Gastroenteritis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Stools
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cases of rotavirus gastroenteritis: Patients will be eligible as cases if they have been identified by the investigator's ongoing rotavirus surveillance studies as having been hospitalized with laboratory-confirmed rotavirus gastroenteritis between January 1, 2007 and June 31, 2009. To be eligible as a case, the child must meet the following criteria: 1) immunocompetent; 2) born after April 15, 2006 (to select a population that would have been in the age group eligible for at least 1 dose of RV5 (RotaTeq); and 3) > 2 months of age on the day of admission.
- Control Subjects: Three controls for each case will be identified using KIDSNET, the state child health registry. Controls will be matched to cases by age and county of residence at birth.

SUMMARY:
The goals of this study are to see what effects the introduction of RV5(RotaTeq) vaccine has had in the community both on the number of rotavirus-associated hospitalizations and on the strains of rotavirus circulating in the community. The investigators will use cases of rotavirus gastroenteritis identified on the wards at Hasbro Children's Hospital during the 2007-2009 rotavirus seasons for a case-control study to estimate rotavirus vaccine effectiveness in preventing rotavirus-associated hospitalizations. The investigators plan to assess rotavirus vaccine coverage in Rhode Island using the state vaccine registry and to examine whether and to what extent rotavirus vaccine was used outside the recommended age limits (off label) during the first 2 years of its implementation in Rhode Island. Finally using the state child health database, KIDSNET the investigators plan to investigate the reasons that children may not have received rotavirus vaccine in order to better target educational efforts for parents and health care providers.

DETAILED DESCRIPTION:
The goals of this study, conducted after the introduction of RV5 (RotaTeq) vaccine in the community, are: 1) to use a case-control study to estimate rotavirus vaccine effectiveness in preventing rotavirus-associated hospitalizations under field conditions, 2) to assess rotavirus vaccine coverage and to examine whether and to what extent rotavirus vaccine was used outside the recommended age limits (off label) during the first 2 years of its implementation in Rhode Island and 3) to investigate risk factors for non-receipt of rotavirus vaccine to inform educational efforts for parents and providers, and 4) to characterize the strains of rotavirus circulating in the community both prior to and after introduction of vaccine to determine if serotype replacement is occurring.

ELIGIBILITY:
Inclusion Criteria:

* rotavirus gastroenteritis requiring hospitalization
* immunocompetent
* born after April 15, 2006
* greater than 2 months of age on the day of admission

Exclusion Criteria:

* rotavirus vaccine contraindicated for that child based on ACIP/AAP recommendations
* an immunization record cannot be obtained through the KIDSNET database

Ages: 2 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Residents of Rhode Island
Sampling Method: Probability Sample
Enrollment: 803 (Actual)
Dates: Start 2009-07 (Actual); Primary Completion 2019-11-01 (Actual); Study Completion 2019-11-01 (Actual)

PRIMARY OUTCOMES:
Rotavirus vaccine effectiveness in preventing rotavirus-associated hospitalizations | 2007-2009
  Rotavirus vaccine effectiveness in preventing rotavirus-associated hospitalizations under field conditions

SECONDARY OUTCOMES:
Vaccine use outside the recommended age limits | 2007-2009
  The extent to which rotavirus vaccine was used outside the recommended age limits (off label) during the first 2 years of its implementation in Rhode Island
Risk factors for non-receipt of rotavirus vaccine | 2007-2009
  Identification of risk factors for non-receipt of rotavirus vaccine
Characterize the strains of rotavirus circulating in the community | 2002-2009
  Characterize the strains of rotavirus circulating in the community both prior to and after introduction of vaccine
Assess rotavirus vaccine coverage | 2007-2009
  Assess rotavirus vaccine coverage in Rhode Island

CONTACTS AND LOCATIONS:
Overall Officials: Penelope H Dennehy, MD, Principal Investigator — Rhode Island Hospital
Locations (1):
- Hasbro Children's Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share IPD since the study uses a deidentified dataset and deidentified stool specimens for serotype analysis